CLINICAL TRIAL: NCT07185880
Title: A Phase 1 Dose Escalation and Randomized Expansion Study of the Safety, Tolerability, and Pharmacokinetics of MT-125 Monotherapy With Radiation in Patients With Newly Diagnosed Glioblastoma
Brief Title: A Phase 1 Study of the Safety and Tolerability of MT-125 in GBM Patients
Acronym: STAR-GBM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Myosin Therapeutics Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MT-125-GBM-101
Record Dates: First submitted 2025-08-19; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma (GBM)
Keywords: Glioblastoma; MGMT unmethylated GBM; IDH wild type; small molecule; MT-125; newly diagnosed; O6-methylguanine- DNA methyltransferase; GBM; isocitrate dehydrogenase (IDH) wild type; non-muscle myosin II
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: This is a FIH, phase 1, open-label, single arm dose escalation study of MT-125. There will be up to 4 dose levels in the dose escalation phase, followed by a dose expansion phase. The dose expansion cohorts will follow a randomized, parallel design with two dose levels determined as the MTD and the dose below the MTD. This study will determine the safety and tolerability of MT-125 administered 5 consecutive days followed by 2 days off per week for the 6 weeks of outpatient RT in participants with newly diagnosed IDH wild-type and MGMT unmethylated GBM. Each dose escalation cohort will enroll no more than 6 total participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MT-125 at 25 mg (Experimental): Up to 6 participants will receive 25 mg of MT-125 for 5 days, then off 2 days for a total of 6 weeks in combination with radiation therapy.
  Interventions: Drug: MT-125
- MT-125 at 50 mg (Experimental): Up to 6 participants will receive 50 mg of MT-125 for 5 days, then off 2 days for a total of 6 weeks in combination with radiation therapy.
  Interventions: Drug: MT-125
- MT-125 at 83.5mg (Experimental): Up to 6 participants will receive 83.5 mg of MT-125 for 5 days, then off 2 days for a total of 6 weeks in combination with radiation therapy.
  Interventions: Drug: MT-125
- MT-125 at 100 mg (Experimental): Up to 6 participants will receive 100 mg of MT-125 for 5 days, then off 2 days for a total of 6 weeks in combination with radiation therapy.
  Interventions: Drug: MT-125
- MT-125 at MTD and one dose lower than MTD (Experimental): Participants will be randomized to receive either MTD or one dose lower than MTD for 5 days, then off 2 days for a total of 6 weeks in combination with radiation therapy.
  Interventions: Drug: MT-125

INTERVENTIONS:
Drug: MT-125 — This is an investigational new drug under IND 170975.

SUMMARY:
The purpose of the study is to determine the recommended dose and further understand the safety of MT-125 in participants who have been diagnosed with glioblastoma, a primary brain tumor, when administered in combination with your standard of care treatment.

Initially, participants with newly diagnosed glioblastoma will be given different doses of MT-125 in combination with radiotherapy (RT) with the goal of identifying the highest tolerated dose.

Up to 36 people with glioblastoma who are at least18 years old are being invited to join this study. MT-125 is a type of study treatment which acts on cancer cells in the brain to destroy them. It will be administered on the same day as your standard of care radiotherapy because it is also designed to help radiotherapy work better. However, this is the first time MT-125 will be studied in humans. Therefore, the use is considered investigational. If you would like more details about MT-125 in glioblastoma participants, please ask the Study Doctor.

You will be among the first participants with glioblastoma to receive this study treatment. Its safety and effectiveness have not yet been established in humans. Thus, we do not know whether it will work for you. Your condition may improve, may get worse, or there may be no change.

The selected participant population-individuals newly diagnosed with histologically and/or molecularly confirmed IDH wild-type, MGMT-unmethylated glioblastoma-represents those least likely to experience safety concerns or adverse events related to the study treatment, and most likely to derive therapeutic benefit.

There are certain tests/questions you must complete to find out if you meet the requirements to be in the study. If you do not meet these requirements, you cannot take part in the study. If this happens, you can talk to your Study Doctor about other options.

DETAILED DESCRIPTION:
MT-125 is a potent, selective, and central nervous system (CNS) permeable dual small molecule inhibitor of the non-muscle myosin II (NMII) paralogs, IIA and IIB. MT-125 is being developed by Myosin Therapeutics Inc. as a potential treatment for glioblastoma (GBM). NMIIs are molecular motor ATPases that act directly on actin to regulate the cytoskeleton's control of cellular processes such as movement, division, signaling and mitochondrial biology. As a result, simultaneous inhibition of NMIIA and IIB with MT-125 interferes with tumor cell proliferation, invasion and metastasis, while also generating reactive oxygen species (ROS) in tumor cells. The latter is due to the role of NMII in mitochondrial quality control and underlies the synergistic survival benefit observed in preclinical studies when MT-125 and radiation therapy (RT) are combined. Additionally, NMIIA is upregulated in several types of cancer, including GBM, speaking to its importance in cancer physiology and making these tumor cells highly sensitive to its inhibition. The focus of this first-in-human (FIH) clinical study is GBM.

Patients with GBM have a poor prognosis, and there have been no new Food and Drug Administration (FDA) approved drugs for these patients since 2008, when bevacizumab was approved. The current well-known standard of care for newly diagnosed GBM is maximal safe surgical resection followed by concurrent RT with temozolomide (TMZ). O6-methylguanine- DNA methyltransferase (MGMT) promoter methylation status is the most predictive biomarker for TMZ responsiveness, where patients with unmethylated MGMT do not respond to TMZ. There is, therefore, an urgent unmet need for effective systemic therapy in patients with unmethylated MGMT.

MT-125 significantly prolongs survival as a monotherapy in animal models and is synergistic with both RT and with FDA-approved oncogenic kinase inhibitors to further enhance survival. In order to develop highly effective combinations of MT-125 with other pharmacologic therapies, we will start with an evaluation of MT-125 as a monotherapy in a first-in-human (FIH) Phase 1 trial with RT in newly diagnosed isocitrate dehydrogenase (IDH) wild type / MGMT unmethylated GBM. In the pivotal 28-day nonclinical safety studies, no dose-limiting toxicities (DLT) or adverse effects (AE) were noted in any of the parameters evaluated (clinical observations, functional endpoints, clinical pathology, macroscopic and histologic tissue assessments) at doses up to the NOAELs, 20 mg/kg/day and 30 mg/kg/day in dogs and rats, respectively, which yielded systemic MT-125 exposures 10- to 16-fold greater than efficacious exposures in pharmacodynamic in vivo models. As the NOAELs in both studies were below the STD10 (rats) and HNSTD (dogs), the calculated safety margins are conservative. Here we will perform a FIH monotherapy trial in newly diagnosed IDH wild type/ MGMT unmethylated GBM with RT.

The goal of this FIH, Phase 1, single arm MT-125 dose escalation study is to evaluate the safety and tolerability of MT-125 administered 5 consecutive days per week with 2 days off for the 6 weeks of outpatient RT. Participants with newly diagnosed GBM with histologically or molecularly confirmed IDH wild type and MGMT unmethylated will be eligible to enroll. We have chosen this subpopulation of patients, as they do not historically benefit from TMZ therapy, which justifies not including treatment with this alkylator in the clinical trial. The DLT observation window will be 6 weeks following first treatment administration, and a Bayesian Optimal Interval (BOIN) trial design will be used to efficiently evaluate up to four dose levels. Secondary endpoints for this Phase 1 study will include determining the maximum tolerated dose (MTD), which will contribute to the selection of the recommended phase 2 dose (RP2D) and evaluating the systemic pharmacokinetics (PK) of MT-125.

Once the MTD is determined, additional participants will be enrolled into a randomized, parallel dose expansion cohort, consisting of up to 2 potential doses of MT-125. The dose levels for the expansion cohort will be selected as the MTD and the dose below the MTD. Overall response rate (ORR) in those participants with measurable disease, progression-free survival (PFS6) in all participants, and Overall Survival (OS) in all participants are included as exploratory endpoints.

If no MTD is identified within the initially defined dose range and all tested doses are deemed well-tolerated based on the observed DLTs, the study may be paused temporarily to allow consideration of dose levels beyond those originally planned.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the informed consent form (ICF).
2. New Diagnosed with histologically or molecularly confirmed IDH wild type and MGMT unmethylated GBM.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2.
4. The following laboratory values obtained ≤15 days prior to registration:

   1. Hemoglobin ≥9.0 g/dL
   2. Absolute neutrophil count (ANC) ≥1500/mm3
   3. Platelet count ≥100,000/mm3
   4. Total bilirubin ≤1.5 x upper limit of normal (ULN)
   5. Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤3 x ULN (or ≤5 x ULN for participants with liver involvement)
   6. Prothrombin time (PT)/ International normalized ratio (INR)/ Activated partial thromboplastin time (aPTT) ≤1.5 x ULN OR if participant is receiving anticoagulant therapy and INR or aPTT is within target range of therapy
   7. Serum eGFR ≥60 ml/min
5. QTc 470 ms on triplicate 12 lead ECG ≤29 days prior to registration. NOTE: QTc intervals will be corrected using Fridericia's formula (Fridericia 1920)
6. Echocardiographic Assessment: Left Ventricular Ejection Fraction (LVEF) ≥ 55%.
7. Negative serum pregnancy test done ≤7 days prior to first dose of MT-125 administration, for persons of childbearing potential only.

   a. If >7 days between last test and first dose of study treatment, the serum pregnancy test will be repeated.
8. Has provided written informed consent.
9. Ability to complete questionnaire(s) by themselves or with assistance.
10. Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
11. On a stable dose of steroids for at least 2 weeks prior to enrollment

Exclusion Criteria:

1. Any of the following because this study involves an investigational agent, the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown:

   1. Pregnant persons
   2. Nursing persons
   3. Persons of childbearing potential and persons able to father a child who are unwilling to employ adequate contraception.
2. Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
3. Receiving any other investigational agent.
4. Any concomitant disease, condition, or treatment that could interfere with the conduct of the study, or that would, in the opinion of the Investigator or Sponsor, pose an unacceptable risk to the participant in the study or interfere with the interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity Measurement | From Day 1 through 6 weeks of treatment
  The dose escalation portion of this study will follow a BOIN design with cohorts containing a min of 3 DLT evaluable participants. If the observed DLT rate at the current dose is ≤0.236, then the decision will be to escalate the dose to the next higher dose level; if the observed DLT rate at the current dose is >0.359, then the decision will be to deescalate the dose to the next lower dose level; otherwise, the decision will be to stay at the current dose level.
Incidence and Severity of AEs | From Day 1 through 6 weeks of treatment
  Incidence and Severity, attribution, grade and type of AE will be assessed based on the NCI CTCAE v5.

SECONDARY OUTCOMES:
Maximum Tolerated Dose | Day 1 through Day 40
  To determine the maximum tolerated dose (MTD) of MT-125
PK Parameters- Cmax | Completed on study days; Day 1, Day 2, Day 5, Day 19, Day 33 and Day 40
  Cmax is the maximum or peak serum concentration at identified timepoints
PK Parameters - Tmax | Completed on study days; Day 1, Day 2, Day 5, Day 19, Day 33 and Day 40
  The time it takes for a drug to reach a maximum concentration after administration
PK Parameters-AUC 0-24hr | Completed on study days; Day 1, Day 2, Day 5, Day 19, Day 33 and Day 40
  Area under the plasma concentration-time curve over the last 24 hour dosing interval
PK Parameters - T1/2 | Completed on study days; Day 1, Day 2, Day 5, Day 19, Day 33 and Day 40
  Time required for plasma concentrations of a drug to decrease by 50%
PK Parameters - CL | Completed on study days; Day 1, Day 2, Day 5, Day 19, Day 33 and Day 40
  CL will quantify the bodies efficiency in eliminating MT-125
PK Parameters - Vss | Completed on study days; Day 1, Day 2, Day 5, Day 19, Day 33 and Day 40
  The steady state volume of distribution that describes how MT-125 distributes throughout the body once it has reached a state of equilibrium
Determine the phase 2 dose | Day 1 through 6 weeks of treatment
  To determine the Recommended Phase 2 Dose (RP2D) of MT-125

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Hegi ME, Genbrugge E, Gorlia T, Stupp R, Gilbert MR, Chinot OL, Nabors LB, Jones G, Van Criekinge W, Straub J, Weller M. MGMT Promoter Methylation Cutoff with Safety Margin for Selecting Glioblastoma Patients into Trials Omitting Temozolomide: A Pooled Analysis of Four Clinical Trials. Clin Cancer Res. 2019 Mar 15;25(6):1809-1816. doi: 10.1158/1078-0432.CCR-18-3181. Epub 2018 Dec 4. PMID 30514777
- [Background] Hegi ME, Diserens AC, Gorlia T, Hamou MF, de Tribolet N, Weller M, Kros JM, Hainfellner JA, Mason W, Mariani L, Bromberg JE, Hau P, Mirimanoff RO, Cairncross JG, Janzer RC, Stupp R. MGMT gene silencing and benefit from temozolomide in glioblastoma. N Engl J Med. 2005 Mar 10;352(10):997-1003. doi: 10.1056/NEJMoa043331. PMID 15758010
- [Background] Melhem JM, Detsky J, Lim-Fat MJ, Perry JR. Updates in IDH-Wildtype Glioblastoma. Neurotherapeutics. 2022 Oct;19(6):1705-1723. doi: 10.1007/s13311-022-01251-6. Epub 2022 May 31. PMID 35641844
- [Background] Kenchappa RS, Radnai L, Young EJ, Zarco N, Lin L, Dovas A, Meyer CT, Haddock A, Hall A, Toth K, Canoll P, Nagaiah NKH, Rumbaugh G, Cameron MD, Kamenecka TM, Griffin PR, Miller CA, Rosenfeld SS. MT-125 inhibits non-muscle myosin IIA and IIB and prolongs survival in glioblastoma. Cell. 2025 Aug 21;188(17):4622-4639.e19. doi: 10.1016/j.cell.2025.05.019. Epub 2025 Jun 10. PMID 40499543
- [Background] Yuan Y, Hess KR, Hilsenbeck SG, Gilbert MR. Bayesian Optimal Interval Design: A Simple and Well-Performing Design for Phase I Oncology Trials. Clin Cancer Res. 2016 Sep 1;22(17):4291-301. doi: 10.1158/1078-0432.CCR-16-0592. Epub 2016 Jul 12. PMID 27407096
- [Background] Liu S, Yuan Y. Bayesian optimal interval designs for phase I clinical trials. Journal of the Royal Statistical Society: Series C (Applied Statistics). 2015;64(3):507-23.